CLINICAL TRIAL: NCT00006478
Title: Pilot Trial to Evaluate Immune Response Using Idiotype Vaccines Following High-Dose Chemotherapy and Hematopoietic Stem Cell Transplantation for Follicular Lymphoma
Brief Title: Vaccine Therapy Following Chemotherapy & Peripheral Stem Cell Transplantation in Treating Non-Hodgkin's Lymphoma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Genitope suspend drug development by decision made by the FDA March 6, 2008.
Sponsor: University of Nebraska (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0260-00-FB; 37-7109-2007-001 (Other Grant/Funding Number: Cattleman's Fund); GENITOPE-IND-8294 (Other Grant/Funding Number: Genitope Corporation)
Record Dates: First submitted 2000-11-06; First posted 2003-01-27 (Estimated); Results first posted 2010-11-17 (Estimated); Last update posted 2023-09-18 (Actual); Status verified 2023-08

CONDITIONS: Lymphoma
Keywords: recurrent grade 1 follicular lymphoma; recurrent grade 2 follicular lymphoma; recurrent grade 3 follicular lymphoma
MeSH Terms: conditions — Lymphoma; Lymphoma, Follicular | interventions — FANG vaccine; keyhole-limpet hemocyanin; sargramostim; Chemotherapy, Adjuvant

ARMS (1):
- Effectiveness of Vaccine Therapy Following Chemotherapy & Peripheral Stem Cell Transplantation (Experimental): Phase II trial to study the effectiveness, safety & toxicity of vaccine therapy following chemotherapy and peripheral stem cell transplantation in treating patients who have non-Hodgkin's lymphoma.
  Vaccinations begin at day 100 or up to 6 months after hematopoietic stem cell transplantation. Participants receive autologous lymphoma-derived idiotype vaccine plus keyhole limpet hemocyanin subcutaneously (SC) on day 1. Sargramostim (GM-CSF) SC is administered on days 1-4. Treatment repeats every 4 weeks for 4 doses, followed 12 weeks later by the fifth and final dose.
  Interventions: Biological: autologous tumor cell vaccine; Biological: keyhole limpet hemocyanin; Biological: sargramostim; Procedure: adjuvant therapy

INTERVENTIONS:
Biological: autologous tumor cell vaccine
Biological: keyhole limpet hemocyanin
Biological: sargramostim
  Other Names: Leukine
Procedure: adjuvant therapy

SUMMARY:
RATIONALE: Vaccines made from a person's cancer cells may make the body build an immune response to kill cancer cells. Vaccine therapy may be an effective treatment for non-Hodgkin's lymphoma.

PURPOSE: Phase II trial to study the effectiveness of vaccine therapy following chemotherapy and peripheral stem cell transplantation in treating patients who have non-Hodgkin's lymphoma.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the humoral and cellular immune responses in patients with follicular non-Hodgkin's lymphoma treated with autologous lymphoma-derived idiotype vaccine with keyhole limpet hemocyanin plus sargramostim (GM-CSF).
* Determine the safety and toxicity of this regimen in these patients in the post-transplant setting.
* Determine the changes in quantitative bcl-2 in the blood and bone marrow of these patients before and at various times after the series of idiotype vaccines.

OUTLINE: Vaccinations begin at day 100 or up to 6 months after hematopoietic stem cell transplantation. Patients receive autologous lymphoma-derived idiotype vaccine plus keyhole limpet hemocyanin subcutaneously (SC) on day 1. Sargramostim (GM-CSF) SC is administered on days 1-4. Treatment repeats every 4 weeks for 4 doses, followed 12 weeks later by the fifth and final dose.

Patients are followed every 3 months for 2 years, every 6 months for 2 years, and then annually thereafter.

PROJECTED ACCRUAL: A total of 20 patients will be accrued for this study.

ELIGIBILITY:
Inclusion Criteria:

* Over 19 years of age
* Histologically proven grade I, II, or III follicular non-Hodgkin's lymphoma that failed induction therapy
* Minimal disease state at day 100 to 6 months post-transplantatio

  * Lymph nodes smaller than 2 centimeters (cm)
  * Less than 20% bone marrow involvement with lymphoma
  * Uncertain complete remission, defined by greater than 75% reduction in the size of the pre-transplantation mass not representing active disease
* Tissue sample safely accessible by biopsy, needle aspiration, or phlebotomy

  o Must have adequate circulating lymphoma cells
* Karnofsky greater than 70%
* Absolute neutrophil count greater than 1,000/mm^3 (No restrictions if study vaccine administered at 6 months after transplantation)
* CD4+ count greater than 200/microliter (No restrictions if study vaccine administered at 6 months after transplantation)
* Bilirubin less than 2.0 mg/dL (unless due to lymphomatous involvement)
* Serum glutamic oxaloacetic transaminase (SGOT) and serum glutamic pyruvic transaminase (SGPT) less than 2 times normal (unless due to lymphomatous involvement)
* Creatinine no greater than 2.0 mg/dL
* Fertile patients must use effective contraception during and for 6 months after study participation

Exclusion Criteria:

* Previously received no more than 2 high-dose chemotherapies before hematopoietic stem cell transplantation
* Not pregnant or nursing/negative pregnancy test

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2000-10-11 (Actual); Primary Completion 2008-04-03 (Actual); Study Completion 2008-04-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Julie M Vose, MD, Study Chair — University of Nebraska
Locations (1):
- University of Nebraska Medical Center, Omaha, Nebraska, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Vaccine Therapy: vaccination to beging at day +100 or 6 months after hematopoietic stem cell transplantation. The vaccine will be given every 4 weeks for 7 consecutive doses and will include Idiotype + KLH along with the adjuvant, GMCSF
Period: Overall Study
Arm/Group | Vaccine Therapy
Started | 19
Completed | 12
Not Completed | 7
Not completed — Vaccine could not be produced | 1
Not completed — Physician Decision | 6

BASELINE CHARACTERISTICS:
Arm/Group | Vaccine Therapy
Number analyzed (Participants) | 19
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 17
  >=65 years | 2
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.7 (10.68)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 9
Region of Enrollment [Number; unit: participants]
  United States | 19

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Humoral and Cellular Immune Response
Description: evaluate the humoral immune responses and cellular immune responses to idiotype vaccine with KLH and GM-CSF adjuvant given to patients with follicular lymphoma following high-dose chemotherapy and autologous stem cell transplantation
Time Frame: immune responses will be obtained prior to first immunization (baseline), prior to the 5th, 6th, 7th immunization series and 2 weeks following administration of the 7th immunization series. And then obtained annually until disease progression
Population: NO formal analysis was completed as this trial was halted prematurely. Thirty patients were to be enrolled in the protocol so that 15 patients would be evaluable at the end of the immunization process. Of the 19 patients enrolled on the trial, only 12 went on to complete the vaccine series.
Arm/Group | Vaccine Therapy
Number analyzed (Participants) | 0

2. Secondary Outcome: Safety of Idiotype Vaccine
Description: To evaluate the safety of idiotype vaccine with KLH and GM-CSF adjuvant in the post-transplant setting
Time Frame: At each immunization and at study completion
Population: The study was terminated early and was not analyzed. At this time, the evaluation of this data is unknown as it has been purged.
Arm/Group | Vaccine Therapy
Number analyzed (Participants) | 0

3. Secondary Outcome: Toxicity of Idiotype Vaccine
Description: To evaluate the toxicity of idiotype vaccine with KLH and GM-CSF adjuvant in the post-transplant setting
Time Frame: At each immunization and at study completion
Population: as for outcome 2
Arm/Group | Vaccine Therapy
Number analyzed (Participants) | 0

4. Secondary Outcome: Changes in Quantitative Bcl-2
Description: To evaluate changes in quantitative bcl-2 of the blood and bone marrow prior to and at various time points following the series of idiotype vaccines.
Time Frame: 1 year post transplant evaluation and then annually until disease progression
Population: as for outcome 2
Arm/Group | Vaccine Therapy
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Description: No serious adverse events were observed. No other (non-serious) adverse event were observed within the reporting threshold.
Arm/Group | Vaccine Therapy
Serious Adverse Events (participants affected / at risk) | 0/19
Other Adverse Events (participants affected / at risk) | 0/19

LIMITATIONS AND CAVEATS:
The Sponsor Genitope suspend development of MyVax in light of the decision made by the FDA March 6, 2008, therefore this trial was halted prematurely leaving insufficient data to analyze.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No